CLINICAL TRIAL: NCT06970769
Title: Comparison of the Effects of Vagus Nerve Stimulation and Breathing Exercise on the Autonomic Nervous System in Mothers of Children With Cerebral Palsy
Brief Title: Effect of Vagus Nerve Stimulation and Breathing Exercise on the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Gamze Demircioğlu, Asst. Prof. Dr., Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-ATLAS-MSEHF-003
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2024-07

CONDITIONS: Mother of a Child With Cerebral Palsy
Keywords: cerebral palsy; mother; autonomic nerve system; vagus; breathing exercises; depression; pain; sleep quality
MeSH Terms: conditions — Cerebral Palsy; Depression; Pain; Sleep Initiation and Maintenance Disorders | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: "vagus nerve stimulation" and "deep breathing exercises." Autonomic nervous system, pain, depression, sleep quality and caregiver burden will be assessed before and after the study.
Who Masked: Participant
Masking Description: This study will employ single masking, where participants will be unaware of their specific group assignment (motor, sensory, or combined motor-sensory exercise groups) to minimize bias. Researchers will know the group assignments to ensure correct administration of interventions, but participants will remain blinded to the type of intervention they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular Nerve Stimulation (Experimental): The auricular branch of the vagus nerve can be superficially stimulated from the external ear by non-invasive access. This method is applied without any surgical procedure by means of TENS add-on devices. This technique, which is widely used in epilepsy, pain and headache, increases the intensity of pain and reduces mechanical sensitivity.
  Interventions: Other: Vagus nerve stimulation
- Deep breathing exercise (Experimental): Deep breathing exercise aimed to improve stress, sleep problems and physiological balance by increasing parasympathetic activity on the autonomic nervous system of mothers in our study. Diaphragmatic breathing technique was taught to participants who applied deep breathing exercise in a comfortable position. Exercises were planned to be performed with a certain rhythm of inspiration and expiration times. Participants were trained with repetitions so that they could continue the application at home. The exercises were applied regularly in the home environment for the specified period.
  Interventions: Other: Deep Breathing Exercises

INTERVENTIONS:
Other: Vagus nerve stimulation — In our study, the auricular branch in the pinna was superficially stimulated with a TENS-based vagustim device for non-invasive vagus nerve stimulation. The application was performed in regular sessions with a physiotherapist according to the recorded protocol. This deactivation aimed at modulation of the autonomic nervous system via the vagus nerve.
  Arms: Auricular Nerve Stimulation
Other: Deep Breathing Exercises — In the study, the participants who were given deep breathing exercises were taught the correct technique in a semi-sitting position. During the exercises, deep breathing and relaxation periods were applied for certain periods. The respiratory rhythm was arranged as controlled inspiration and expiration. The participants were given an application practice so that they could continue the exercise at home.
  Arms: Deep breathing exercise

SUMMARY:
This project will compare the effects of intraaural vagus nerve stimulation and deep breathing exercises on the autonomic nervous system in mothers of children with cerebral palsy. This approach will allow researchers to evaluate the effects of these practices on the autonomic nervous system.

The study is planned to include 38 mothers of children with cerebral palsy between the ages of 18-50. Participants will be informed about the purpose of the study and will provide written informed consent to verify voluntary participation. Participants will be randomly assigned to one of two groups: "vagus nerve stimulation" and "deep breathing exercises." Autonomic nervous system, pain, depression, sleep quality, and caregiver burden will be assessed before and after the study.

DETAILED DESCRIPTION:
The autonomic nervous system plays an important role in maintaining the physiological and psychological balance of individuals. Therefore, irregularities in the autonomic nervous system can negatively affect daily life activities and quality of life. In mothers of children with cerebral palsy, the stress, sleep problems and physical loads brought about by the caregiving process can disrupt the autonomic nervous system functions. In this context, interventions aimed at supporting autonomic balance are gaining importance. This project will compare the effectiveness of intraaural vagus nerve stimulation and deep breathing exercises used in clinical settings on the autonomic nervous system in healthy individuals and will allow researchers to evaluate the effects of these methods on physiological functions.

The study plans to include 38 mothers of children with cerebral palsy between the ages of 18-50. Participants will be informed about the purpose of the study and will provide written informed consent to confirm voluntary participation. Participants will be randomly assigned to one of two groups: "vagus nerve stimulation" and "deep breathing exercises." Autonomic nervous system, pain, depression, sleep quality and caregiver burden will be assessed before and after the study. Data analysis was performed using SPSS v.26 (SPSS Inc., USA) software. χ² test was applied in the analysis of qualitative variables. For data that did not show a normal distribution or were ordinal, Wilcoxon test was preferred for within-group comparisons, and Mann-Whitney U test was preferred for between-group comparisons. For numerical data that showed a normal distribution, Paired Samples T-Test was used for within-group comparisons, and Independent Samples T-Test was used for between-group comparisons. Effect size values were classified as 'negligible' in the range of 0-0.19, 'small' in the range of 0.20-0.49, 'medium' in the range of 0.50-0.79, and 'large' in the range of 0.80 and above. The significance level was determined as p<0.05 in all statistical tests performed.

ELIGIBILITY:
Inclusion Criteria:

* Having a child diagnosed with cerebral palsy
* The child must be between 4-18 years old
* The mother must be between 18-50 years old
* The mother to be studied must be literate

Exclusion Criteria:

* Providing care for an elderly, chronically ill or disabled relative;
* Having a history of chronic disease such as diabetes, cardiovascular or pulmonary disease, kidney disease, musculoskeletal disorders or any psychiatric disorder
* Caring for another child under the age of two
* Having another child at home who needs special health care
* Not volunteering to participate in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Gross motor functional classification (GMFCS) | Baseline (prior to intervention)
  It can be found by palisino for the operation of gross motor function in children with cerebral palsy, it is a scale with proven validity and reliability. It is specially prepared for children with cerebral palsy up to 12 years of age, depending on the independence and independent movements allowed in movements such as transfer and mobilization, the limitation in functionality and the use of assistive devices. age, 12-15 years, 15-18 years). The GMFCS categorizes motor function into five levels (I to V), where Level I indicates the highest level of independence and functional ability, and Level V represents the most severe motor limitations. Therefore, higher levels correspond to poorer outcomes in terms of gross motor function.
beck depression scale | 3 week
  The Turkish version of the Beck Depression Scale, which has been validated and reliable in Turkish, was used to assess depression. Each question is scored between 0-3 and consists of 4 items. The survey consists of 21 questions. The total score is calculated as 63 points by evaluating symptoms and behavior. The scale includes; pessimism, sleep disorders, self-hatred, mood, desire to punish oneself, dissatisfaction, guilt, sense of failure, sense of punishment, somatic disorder, exhaustion, fatigue, body perception status change, self-blame, crying spells, determination of workability, stress, social isolation, difficulty in decision making, eating status, weight loss and sexual issues. The higher the final score of the survey, the higher the level of depression. According to the scale scores; 0-9 is interpreted as "no or minimal depression", 10-16 as "mild depression", 17-29 as "moderate depression", and 30-63 points as "severe depression".
Caregiving Burden Scale | 3 week
  The Caregiving Burden Scale, developed to assess the perceived burden in caregivers, was created by Zarit and his colleagues in 1980. The Turkish validity and reliability study was conducted by İnci and Erdem. The scale is a 22-item, 5-point Likert-type scale that measures the social and emotional difficulties experienced during the care process. Each item is scored between 0-4, and the total score ranges from 0 to 88. As the score increases, the perceived care burden increases proportionally. According to the evaluation results; 0-20 is considered low or almost no burden, 21-40 is considered mild-moderate burden, 41-60 is considered moderate-high burden, and 61-88 is considered excessive burden. In the reliability study of the Turkish form, the Cronbach Alpha coefficient was determined as 0.95, and the test-retest reliability was found to be 0.90. In addition, according to factor analysis, the scale has a one-dimensional structure and effectively reflects the stress level.
NORDIC musculoskeletal system questionnaire | 3 week
  The Scandinavian Musculoskeletal System Questionnaire was employed to identify painful regions in the participants. This tool evaluates musculoskeletal complaints in areas such as the lower back, neck, shoulders, and other body regions. It offers reliable information regarding the onset, prevalence, and consequences of symptoms experienced over the past 12 months and the previous 7 days across nine categorized anatomical regions (feet/ankles, knees, thighs, hips, hands/wrists, lower back, elbows, upper back, shoulders, and neck). The questionnaire can be completed independently or through an interviewer-administered format. The NMQ-E records the presence of symptoms in each region using binary (yes/no) responses, and results are reported as percentages. Higher percentages indicate a greater prevalence of musculoskeletal complaints in the corresponding region, reflecting poorer outcomes.
Pittsburgh Sleep Quality Index (PSQI) | 3 week
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess the sleep quality of the participants. It is a questionnaire that evaluates sleep quality and current sleep disorders within a one-month period. The PSQI consists of 19 items and is scored under 7 components. These components are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleeping pills, and daytime dysfunction. The participant obtains a general sleep quality score by summing the scores from the seven components . Apart from these components, there are 5 additional questions in the rest of the questionnaire that must be answered by the participant's bed partner if the participant has one. However, these 5 questions are not used in the total score, but are used in clinical interpretation . All 19 questions are scored between 0 and 3. A score of 0 for each component indicates that there is no difficulty with that question, while a score of 3 indicates t
Autonomic Nervous System Assessment (Polar H10) | 3 week
  The Polar H10 device is a reliable and sensitive sensor that evaluates autonomic nervous system (ANS) functions via heart rate variability (HRV). In the Cubios system, multiple HRV parameters-including HR (bpm), RMSSD (ms), SDNN (ms), LF (ms²), and HF (ms²)-are integrated into a single analytical model to assess overall autonomic nervous system (ANS) function. Although each parameter has a different measurement unit, the system processes them collectively to produce a unified outcome. Therefore, these measures are not reported individually but are synthesized into a composite ANS balance evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Atlas University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this study. All collected data will be used solely for the purpose of analyzing study outcomes and will remain confidential. This approach is taken to ensure the privacy and confidentiality of participant information.